CLINICAL TRIAL: NCT03909620
Title: A Study Assessing the Utility of Low-dose Computed Tomography (LDCT) in Lung Cancer Screening in North India
Brief Title: Utility of LDCT in Lung Cancer Screening in a TB Endemic Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Navneet Singh, Additional Professor, Department of Pulmonary Medicine, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NK/5292/DM/760
Record Dates: First submitted 2019-04-05; First posted 2019-04-10 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Lung Cancer
Keywords: lung cancer; ldct; low-dose CT; screening; lung nodule
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDCT arm (Experimental): All eligible participants will undergo screening with LDCT
  Interventions: Diagnostic Test: Low-dose computed tomography of chest

INTERVENTIONS:
Diagnostic Test: Low-dose computed tomography of chest — Eligible subjects will undergo a single round of LDCT screening. The LDCT will be considered as positive if a solid nodule or part-solid nodule of size ≥6 mm or non-solid nodule of size ≥20 mm is identified. Evaluation of positive nodules will be performed as per existing standard recommendations
  Other Names: LDCT; Low-dose CT

SUMMARY:
Lung cancer screening with low-dose computed tomography (LDCT) has been recently shown to result in a significant reduction in lung cancer-specific mortality. However, the utility of LDCT screening in developing countries with high incidence of tuberculosis has not been adequately studied. The investigators hypothesize that LDCT screening in tuberculosis endemic regions is likely to yield a large proportion of false-positive results, especially in the initial round of screening, posing a significant burden on the healthcare system. Herein, the investigators assess the utility of LDCT and its cost-effectiveness in India.

DETAILED DESCRIPTION:
Screening for lung cancer may reduce lung cancer mortality by diagnosing the disease at an early stage when it is treatable more effectively. There are several methods available for screening of lung cancer. These include sputum cytology, chest radiography, computed tomography (CT) of the chest, and positron emission tomography (PET). However, sputum cytology and chest radiography have been found to be ineffective as screening tests for lung cancer as there is no reduction in lung cancer mortality. The use of CT or PET for lung cancer screening may be associated with unacceptable levels of radiation exposure and enormous cost.

Low-dose computed tomography (LDCT) of the chest is a special type of CT, which uses relatively low radiation exposure to create a low-resolution image of the entire thorax. The radiation exposure associated with LDCT is 5-6 times less than that of a conventional CT scan of the thorax. LDCT screening has been to shown to result in a 20% reduction in lung cancer-specific mortality. Several national and international guidelines recommend this strategy for lung cancer screening.

Despite these guidelines and recommendations by several organizations, lung cancer screening has not been established in several developing countries, where a controversy arises due to high rates of granulomatous diseases like tuberculosis. Emerging evidence indicates that false positive results with LDCT in developing countries may not be unacceptably high as previously believed.

In this study, the investigators intend to assess the utility of lung cancer screening using low-dose computed tomography (LDCT) in India, a country with high prevalence of tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 55-74 years with at least 30 pack-year history of smoking (or smoking index ≥600) who are current smokers or quit within the last 15 years OR
* Individuals aged 50-74 years with at least 20 pack-year history of smoking (or smoking index ≥400) who are current or former smokers with COPD or family history of lung cancer in any first-degree relative

Exclusion Criteria:

* Symptomatic structural lung disease other than COPD (e.g. bronchiectasis, chronic pulmonary aspergillosis, pulmonary fibrosis)
* Severe comorbid condition which is likely to limit the survival of the patient in the opinion of the investigator (e.g. advanced lung disease, cardiovascular disease, chronic kidney disease, chronic liver disease)
* Presence of symptoms which lead to a suspicion of lung cancer (e.g. hemoptysis or unexplained weight loss [>5 kg] within the last 6 months)
* Conditions which may interfere interpretation of CT (e.g. metallic implants on chest wall, cardiac pacemakers)
* Treatment for any other cancer in the last 5 years
* Pulmonary infection (for which treatment with antimicrobials is indicated) which is active at present or was recent (within the last 3 months)
* Patients who have underwent CT chest within the last 18 months
* Negative consent

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Positivity rate with LDCT screening | After baseline LDCT scan results are available (an average of 1 week after LDCT scan)
  The proportion of participants with a positive result among the total number of individuals screened with LDCT

SECONDARY OUTCOMES:
Rate of detection of lung cancer | Up to 6 months after the LDCT scan
  Rate of lung cancer detection among study participants
False positive rate | Up to 6 months after the LDCT scan
  Rate of false positive results with LDCT screening
Proportion of patients requiring additional procedures (imaging/invasive procedures) | Up to 6 months after the LDCT scan
  The proportion of patients with positive results on initial LDCT scan requiring additional procedures (imaging/invasive procedures)
Proportion of patients developing complications due to additional procedures | Up to 2 weeks after the diagnostic procedure
  The proportion of patients among those who developed complications due to additional procedures (imaging/invasive procedures) performed after initial LDCT scan
Change in the 6-item Spielberger State-Trait Anxiety Inventory (STAI-6) questionnaire score | After communication of baseline LDCT results (an average of 1-2 weeks after the LDCT scan)
  Change in anxiety levels from baseline after conveying LDCT results to the patient
Cost in Indian Rupees to detect one case of lung cancer by LDCT screening | Up to 6 months after the LDCT scan
  Cost-effectiveness of LDCT screening
Proportion of patients who quit/re-initiated smoking after inclusion in study | Up to 6 months after the LDCT scan
  The proportion of patients who quit/re-initiated smoking after inclusion in study

CONTACTS AND LOCATIONS:
Overall Officials: Kuruswamy T Prasad, MD, DM, Principal Investigator — Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh; Rajinder Basher, MD, Principal Investigator — Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh; Mandeep Garg, MD, Principal Investigator — Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh; Sandeep Grover, MD, Principal Investigator — Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh; Naveen Kalra, MD, Principal Investigator — Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh; Navneet Singh, MD, Principal Investigator — Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh; Kathirvel Soundappan, MD, Principal Investigator — Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh, India

IPD SHARING:
Plan to Share IPD: No